CLINICAL TRIAL: NCT06214351
Title: Mobile Midwifery Application: the Effect of Mobile Midwifery Care Provided During the Prenatal Period on Pregnant Women's Stress, Fear of Birth, Preparation for Birth, and Satisfaction with Care
Brief Title: Mobile Midwifery Application Offered in the Prenatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Rumeysa Taskin, Lecturer, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Atatürk Uni.
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Mobile Application
Keywords: Midwife; Prenatal period; Mobile application; Fear of birth; Midwifery care; Readiness

STUDY DESIGN:
Intervention Model Description: Mobile midwifery application is a mobile application based on the prenatal process, where pregnant women can get information about pregnancy, birth and postpartum processes.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): A mobile application will be installed on the smartphones of the pregnant women in the experimental group.
  The mobile application will be installed on the phones of the pregnant women in the experimental group. (The mobile application will be downloaded from the "Play Store" for Android users and from the "App Store" for iOS users). Information about the application will be provided and any questions from the pregnant women will be answered. Pregnant women will be free to access the application at any time during the study.
  Interventions: Other: Use of mobile midwifery application
- Control Group: (No Intervention): Pregnant women in the control group will receive routine antenatal care. Routine antenatal care will be provided to pregnant women in the control group.

INTERVENTIONS:
Other: Use of mobile midwifery application — Pregnant women in the experimental group will have a mobile midwifery application installed on their smartphones. The pregnant woman will be able to reach the research midwife 24/7. With the informative content and algorithm mechanism in the application, she will be able to provide individual care and detect early signs of danger, enabling her to seek medical attention.
  Arms: Experimental Group

SUMMARY:
In this study, the development of a mobile application for prenatal midwifery care and the examination of the effect of the developed mobile application on the stress, fear of childbirth, readiness for childbirth, and satisfaction with care of pregnant women are aimed. The research has a randomized controlled experimental design. Research data will be collected between January 2024 and October 2024 at the Obstetrics and Gynecology Clinic of Ağrı Training and Research Hospital. The universe of the research will consist of pregnant women who apply to the NST unit and Obstetrics and Gynecology Clinic of the relevant hospital. The sample of the research consists of pregnant women who meet the inclusion criteria and volunteer to participate in the research. A priori power analysis was conducted to determine the sample size of the research. Cohen's standardized effect size reference method was selected in the power analysis. It was calculated that 102 pregnant women (Experimental group: 51, Control group: 51) should be included in order to achieve 80% power with a 95% confidence interval at a significance level of 0.05. In order to account for possible data losses, it was decided to collect data from a total of 128 individuals by including an additional 25% reserve sample in this number. The sample of the research will be selected by randomization among those who meet the specified research criteria. The assignment of participants to the experimental and control groups will be done through randomization. For randomization, the Random Integer Generator method in the Numbers subheading of the https://www.random.org site will be used to create single-group columns between 1 and 128 in the system. In the data collection stage of the study, an Introductory Information Form, Risk Assessment Form of the Ministry of Health of the Republic of Turkey, Visual Analog Patient Satisfaction Scale, Tilburg Pregnancy Distress Scale, Prenatal Self-Evaluation Scale - Fear of Childbirth and Sub-dimensions of Readiness for Childbirth, and Mobile Application Evaluation Form will be used.

DETAILED DESCRIPTION:
Experimental Group: Pregnant women in the experimental group will have a mobile application installed on their smartphones.

Control Group: Pregnant women in the control group will receive routine antenatal care.

Pregnant women who meet the inclusion criteria of the study will be provided with information about the purpose, content, and application of the study. Pregnant women in the experimental and control groups will be included in the study. At this stage, both groups will fill out the Personal Information Form, the Birth Fear and Birth Readiness sub-scales of the Prenatal Self-Evaluation Scale, the Tilburg Pregnancy Distress Scale, and the Risk Assessment Form of the Ministry of Health of the Republic of Turkey.

At the end of the information process, informed consent will be obtained from pregnant women. Pregnant women will be assigned to experimental and control groups using a simple random table from the www.random.org website.

In the last trimester of pregnancy (weeks 38-40), the Birth Fear and Readiness sub-scales of the Prenatal Self-Assessment Scale, Visual Analog Patient Satisfaction Scale, and Tilburg Pregnancy Distress Scale will be administered to both the control and experimental groups. Pregnant women in the experimental group will also complete the mobile application evaluation form.

ELIGIBILITY:
Inclusion Criteria:

Being literate Being 18 years or older Being primigravida Having a single fetus Being in the first and second trimester of pregnancy Having a smartphone and having the ability to use it effectively Having internet access Being open to communication Not having a diagnosed psychiatric disease Volunteering to participate in research

Exclusion Criteria:

Being illiterate Being multiparous Having a High Risk Pregnancy according to the "Risk Assessment Form" of the Ministry of Health of the Republic of Turkey Having a diagnosed psychiatric disorder don't have a disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 and over, pregnant
Enrollment: 107 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Patient Satisfaction Scale | It will be taken at 38-40 weeks of pregnancy.
  The patient satisfaction scale was designed to measure the patient's satisfaction with the given care practices. The scale has numbers from 1 to 10 on a vertical line. Number 1 symbolizes complete dissatisfaction and number 10 symbolizes high level of satisfaction.
Tilburg Pregnancy Distress Scale | This form will be collected at the first meeting with the pregnant woman and at 38-40 weeks of pregnancy.
  It is used to determine distress (stress, anxiety, depression) during pregnancy. The scale consists of a total of 16 items. Each item of the scale is rated as a 4-point Likert type ranging from "very often" (0 points), "quite often" (1 point), "occasionally" (2 points), "rarely or never" (3 points). A total score of 28 or above from the scale enables the diagnosis of pregnant women who are at risk for distress (depression, anxiety, stress).
Prenatal Self-Assessment Scale- Fear of Birth and Birth Readiness Sub-Dimensions | This form will be collected at the first meeting with the pregnant woman and at 38-40 weeks of pregnancy.
  The scale is used to evaluate the adaptation of pregnant women to pregnancy and motherhood. The "Fear of Birth" and "Readiness for Birth" subscales in the scale will be used. Items are evaluated with scores ranging from "1" to "4" (4: "Describes very much," 3: "Partly describes," 2: "Somewhat describes," 1: Does not describe at all"). The lowest score to be taken separately in the fear of birth and birth readiness sub-dimensions is 10 and the highest score is 40.
Mobile Application Evaluation Form | The questionnaire will be filled out for pregnant women in the experimental group at the end of the study (38-40 weeks of pregnancy).
  This is an evaluation form consisting of 8 questions by which pregnant women participating in the study can evaluate the application.
Risk Assessment Form of the Ministry of Health of the Republic of Turkey | It will be filled in at the first meeting with the pregnant woman.
  With this form, it will be determined whether the pregnant women who will participate in the study are at high risk. Pregnant women in the high risk group will not be included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla KANBUR, Principal Investigator — Ataturk University
Locations (1):
- AgriIbrahimCecenU, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No